CLINICAL TRIAL: NCT03817411
Title: A Phase II Randomized Trial of Telatinib in Combination With Capecitabine/Oxaliplatin Versus Capecitabine/Oxaliplatin as First-Line Therapy in Patients With HER2-negative Advanced Adenocarcinoma of the Stomach or Gastroesophageal Junction
Brief Title: Telatinib in Combination With Capecitabine/ Oxaliplatin in 1st Line Gastric or GEJ Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou EOC Pharma Co., Ltd. (Industry)
Collaborators: Shanghai East Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EOC315B2101
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — telatinib; Capecitabine; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telatinib+Capecitabine+Oxaliplatin (Active Comparator): Patients receive Telatinib orally (PO) twice daily (bid) on days 1-21 and Capecitabine PO on days 1-14, then stopped for 7 days, and Oxaliplatin by intravenous injection on day 1 of every cycle. Courses repeat every 21 days.
  Interventions: Drug: Telatinib; Drug: Capecitabine; Drug: Oxaliplatin
- Placebos+Capecitabine+Oxaliplatin (Placebo Comparator): Patients receive placebo orally (PO) twice daily (bid) on days 1-21 and Capecitabine PO on days 1-14, then stopped for 7 days, and Oxaliplatin by intravenous injection on day 1 of every cycle. Courses repeat every 21 days.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Placebos

INTERVENTIONS:
Drug: Telatinib — 300 mg tablets, 900 mg twice daily (BID) at 12h-intervals.
  Other Names: EOC315
  Arms: Telatinib+Capecitabine+Oxaliplatin
Drug: Capecitabine — 1000 mg/m²,twice daily for 14 days followed by a 7-day rest period (14 days on/7 days off schedule).
Drug: Oxaliplatin — 130 mg/m2, administered intravenously over 2 hours, on Day 1 every 3 weeks (one administration per cycle) for a maximum of 6 cycles.
Drug: Placebos — 300 mg tablets, 900 mg twice daily (BID) at 12h-intervals.
  Arms: Placebos+Capecitabine+Oxaliplatin

SUMMARY:
The purpose of the trial is to compare the combination regimen of Telatinib and Capecitabine and Oxaliplatin vs. Capecitabine and Oxaplatin to explore superiority of the Telatinib combination in terms of progression-free survival (PFS) in patients previously untreated for advanced HER2 negative advanced gastric or Gastroesophageal Junction adenocarcinoma.

DETAILED DESCRIPTION:
This trial is a Phase 2, prospective, double-blind, randomized, comparative, multicenter trial in patients with advanced HER2 negative adenocarcinoma of the stomach or Gastroesophageal Junction which has progressed after resection and adjuvant or neoadjuvant therapy, or is unresectable or metastatic at time of first diagnosis. a total of approximately 90 patients will be enrolled and randomized into Telatinib combined with Capecitabine and Oxaliplatin or chemotherapy combined with placebo. All patients will be treated until progressive disease (radiologically documented or symptomatic deterioration) or the occurrence of unacceptable toxicity, withdrawal of consent or investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 and <75 years old at the time of screening.
2. Histologically or cytologically confirmed unresectable locally advanced or metastatic HER2 negative (or HER2 status unknown), gastric or gastro-oesophageal junction adenocarcinoma.
3. Measurable or evaluable lesion as defined by RECIST v1.1.
4. No prior treatment for advanced disease. Adjuvant or neoadjuvant chemotherapy must be stopped at least for 6 months.
5. Prior surgery and/or radiotherapy stopped for at least 4 weeks.
6. ECOG Performance Status 0-1.
7. Life expectancy of at least 3 months.
8. Adequate bone marrow function as evidenced by meeting all of the following requirements:

   1. Absolute neutrophil count > 1.5 × 10 E+9/L without the use of hematopoietic growth factors
   2. Platelet count > 90 ×10 E+9/L without the need for transfusion in the 2 weeks prior the first dose
   3. Hemoglobin >90 g/L without the need for transfusion in the 2 weeks prior the first dose
9. Adequate hepatic function as evidenced by meeting all of the following requirements:

   1. Serum total bilirubin ≤1.5 x upper limit of normal (ULN) (biliary drainage is allowed for biliary obstruction)
   2. Serum albumin levels ≥3.0 g/dL
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) and and alkaline phosphatase (ALP): ≤3.0 x upper limit of normal (ULN) (≤5 x ULN if liver metastases are present and if liver and/or bone metastases ALP ≤ 5 × ULN.)
10. Adequate renal function as evidenced by

    1. serum creatinine ≤1.5 x ULN and creatinine clearance of ≥50 mL/min (Cockcroft-Gault formula).
    2. Urine dipstick for proteinuria of less than 2+ (other ways of urinalysis are also acceptable); if urine dipstick is ≥ 2+, proteinuria must be < 2 g in 24 hours.
11. Prothrombin time (PT) or activated partial thromboplastin time (APTT) and International Normalized Ratio (INR) ≤1.5 x ULN.
12. Recovered from the effects of any prior surgery, radiotherapy or other anti-neoplastic adjuvant therapy. Unresolved toxicity > Grade 1 (except alopecia) from previous anticancer therapy (including radiotherapy) is accepted
13. If female of childbearing potential, the patient must present with a negative urine pregnancy test and agrees to employ adequate birth control measures for at least 90 days after the duration of the study
14. Male who are not sterile agrees to take effective contraception for at least 90 days after the last dose of drug and avoid donating sperm at the same time period.
15. Ability to swallow pills and no major intestinal surgery.
16. Able to understand and sign an informed consent

Exclusion Criteria:

1. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg).
2. Active and uncontrolled central nervous system (CNS) metastases .
3. During the screening and study period, standard dose of anticoagulant or thrombolytic drugs are used for treatment;
4. History of any second malignancy in the last 5 years; patients with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they have been continuously disease free for at least 5 years.
5. Evidence of tumor invasion of major blood vessels by images(including complete proximity, surrounding or extending into the main vascular lumen, such as the pulmonary artery or the superior vena cava), and the investigator judged that it was not suitable for enrollment.
6. A significant thrombotic or hemorrhagic event ≤ 6 months prior to Screening (includes hemoptysis, gastrointestinal bleeding, hematemesis, CNS hemorrhage, severe epistaxis or vaginal bleeding, cerebral infarction, transient ischemic attacks, myocardial infarction, angina, and uncontrolled coronary artery disease).
7. History of active gastroduodenal ulcer, abdominal fistula as well as nongastrointestinal fistula, gastrointestinal perforation or intraabdominal abscess within 6 months prior to screening.
8. Significant cardiac conduction abnormalities, including a history of long QTc syndrome and/or pacemaker.New York Heart Association Class III or IV congestive heart failure, ventricular arrhythmias
9. Exposure to any other investigational or commercial anticancer agents or therapies (Chinese herbal medicines e.g) administered with the intention to treat malignancy within 28 days.
10. Active infection or an unexplained fever during screening visits or on the first scheduled day of dosing (at the discretion of the Investigator, patients with tumor fever may be enrolled), which in the investigator's opinion might compromise the patient's participation in the trial or affect the trial outcome.
11. Positive test or known history of for human immunodeficiency virus (HIV), active hepatitis B (HBsAg) or hepatitis C (anti-HCV antibody) or syphilis (syphilis antibody)
12. If female, the patient is pregnant or lactating at the time of enrollment.
13. Known hypersensitivity to any of the components of fluoropyrimidines or platinum cmpounds.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2021-01-25 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  the proportion of patients with complete response (CR) or partial response (PR) among all patients assessed per RESIST v1.1.

SECONDARY OUTCOMES:
PFS | 24 months
  Progression free survival of All the Evaluable Participants.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of diameters of target lesions, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
CBR | 24 months
  Clinical Benefit Rate, defined as CR+PR+SD≥ 24 weeks
DCR | 24 months
  the proportion of patients who had a best response rating of complete response, partial response, or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D., Study Chair — Shanghai Easter Hospital, Dpt. of Clinical Oncology; Tian Shu Liu, M.D., Study Chair — Shanghai Fudan Zhongshan Hospital, Dpt. of Clinical Oncology
Locations (1):
- Shanghai Easter Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided